CLINICAL TRIAL: NCT01726270
Title: A 8-week, Open-label, Uncontrolled, Exploratory Actual Use Study of Tamsulosin 0.4mg in Men With Prostate Urinary Symptoms in a Simulated Over-the-Counter Environment
Brief Title: An 8-week, Open-label, Uncontrolled Study of Tamsulosin 0.4mg in Men With Bothersome Urinary Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 527.82
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tamsulosin

ARMS (1):
- tamsulosin hydrochloride (Experimental): patients will take drug for 8 weeks in this exploratory study
  Interventions: Drug: tamsulosin

INTERVENTIONS:
Drug: tamsulosin — 0.4 mg

SUMMARY:
Multicenter trial conducted in Pharmacy retail centers

ELIGIBILITY:
Inclusion criteria:

1. Men 18 years of age and older.
2. Able to speak, read and understand English.
3. Willing to participate in the study and voluntarily sign an informed consent document.

Exclusion criteria:

1. Subject or anyone in their household is currently employed by a marketing or marketing research company, and advertising agency or public relations firm, a pharmacy or pharmaceutical company, a manufacturer of medicines, a managed care or health insurance company as a healthcare professional or healthcare practice.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- United States (18):
  - Boehringer Ingelheim Investigational Site, Hoover, Alabama
  - Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - Boehringer Ingelheim Investigational Site, Encino, California
  - Boehringer Ingelheim Investigational Site, Garden Grove, California
  - Boehringer Ingelheim Investigational Site, La Habra, California
  - Boehringer Ingelheim Investigational Site, Anoka, Minnesota
  - Boehringer Ingelheim Investigational Site, Elk River, Minnesota
  - Boehringer Ingelheim Investigational Site, Fridley, Minnesota
  - Boehringer Ingelheim Investigational Site, Roseville, Minnesota
  - Boehringer Ingelheim Investigational Site, Saint Francis, Minnesota
  - Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - Boehringer Ingelheim Investigational Site, Longview, Texas
  - Boehringer Ingelheim Investigational Site, Tyler, Texas
  - Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - Boehringer Ingelheim Investigational Site, Layton, Utah
  - Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - Boehringer Ingelheim Investigational Site, Syracuse, Utah
  - Boehringer Ingelheim Investigational Site, Richmond, Virginia

REFERENCES:
- [Derived] Roehrborn CG, Lowe FC, Gittelman M, Wruck JM, Verbeek AE. Management of Male Lower Urinary Tract Symptoms in a Simulated, Over-the-Counter Setting: An Exploratory Study of Tamsulosin. Drugs Aging. 2019 Feb;36(2):179-188. doi: 10.1007/s40266-018-0621-8. PMID 30607798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 parts: In part 1 participants reviewed the product label and responded to a question about whether the product is appropriate for them to use (self-selection), selected participants then entered part 2 where they recieved study product (actual use).
Groups:
- All Subjects: Part 1 included subjects who answer the self-selection question, probing question and follow-up questions.
  Part 2 included subjects who self-selected to use the product, purchase the product and took at least one dose of drug and participate in at least 1 phone interview.
Period: Part 1, Self-Selection Phase
Arm/Group | All Subjects
Started | 689
Completed | 679
Not Completed | 10
Not completed — Withdrawal by Subject | 10
Period: Eligibility for Part 2
Arm/Group | All Subjects
Started | 389 (No. of subjects potentially eligible for Part 2)
Completed | 369
Not Completed | 20
Not completed — Eligible but did not enter Part 2 | 20
Period: Part 2, Actual-Use Phase
Arm/Group | All Subjects
Started | 369 (20 subjects were eligible for Part 2 but did not enter Part 2)
Completed | 330
Not Completed | 39
Not completed — Withdrawal by Subject | 21
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 5
Not completed — Other than reason specified above | 7

BASELINE CHARACTERISTICS:
Population: Evaluable Analysis Set for Self-Selection (Eval-SS): All subjects who answered self-selection question, probing question and follow-up questions
Arm/Group | All Subjects
Number analyzed (Participants) | 679
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 679

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Appropriately Followed the Label Instructions
Description: Includes subjects who reported:
  1. No improvement in urinary symptoms and stopped taking product,
  2. Reported worsening of urinary symptoms and stopped taking the product,
  3. Reported a new urinary symptom and stopped taking the product,
  4. Reported no "Stop Use" condition and never took more than 1 capsule on any given day,
  5. Reported a "Stop Use" condition and contacted a provider.
Time Frame: 8 weeks
Population: Full Analysis Set for Actual Use Study (FAS-AUS), all subjects who self-selected to use the product, purchased the product, took at least one dose of the product and participated in at least one phone interview.
Measure: Number; unit: Percentage of participants
Groups:
- Tamsulosin Hydrochloride: Participants received tamsulosin hydrochloride 0.4mg capsules, orally, for 8 weeks.
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 321
Percentage of participants | 85.4

2. Secondary Outcome: Percentage of Participants Who Took no More Than One Capsule Per Day
Description: Percentage of participants who took no more than one capsule per day
Time Frame: 8 weeks
Population: Subjects who completed all three telephone follow-up interviews out of the FAS population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 300
Percentage of participants | 93.7 [90.3 to 96.1]

3. Secondary Outcome: Percentage of "Use-Days" for All Participants Who Took no More Than One Capsule Per Day
Description: "Use-day" was defind as a calendar day for which data were available regarding use or non-use.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 321
Percentage of participants | 94.1 [90.9 to 96.2]

4. Secondary Outcome: Percentage of Participants < 45 Years of Age Who Spoke to a Doctor During the Actual Use Phase
Description: Includes participants who:
  1. were less than 45 years of age at enrollment, and
  2. spoke to a doctor during the actual use phase.
Time Frame: 8 weeks
Population: Full Analysis Set for Actual Use Study- Under 45 years (FAS-AUS45), all subjects less than 45 years of age who self-selected to use the product, purchased the product, took at least one dose of the product and participated in at least one phone interview
Measure: Number; unit: Percentage of participants
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 23
Percentage of participants | 30.4

5. Secondary Outcome: Percentage of Participants Who Are Potentially at Risk of Harm by Incorrectly Selecting to Use the Study Product Out of the Total Study Population
Description: Percentage of participants who are potentially at risk of harm by incorrectly selecting to use the study product out of the total study population
Time Frame: 8 weeks
Population: Evaluable Analysis Set for Self-Selection (EVAL-SS), all subjects who answered the self-selection question, probing question and followup questions.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 679
Percentage of participants | 20.9 [17.9 to 24.2]

6. Secondary Outcome: Percentage of Participants Who Have a Correct Self-selection Response Out of the Total Study Population
Description: Percentage of participants who have a correct self-selection response as defined by the "Uses", "Allergy alert", and "Do Not Use" sections of the Drug Facts Label.
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamsulosin Hydrochloride
Number analyzed (Participants) | 679
Percentage of participants | 73.9 [70.5 to 77.2]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Treated set
Groups:
- EVAL-SS: Evaluable Analysis Set for Self-Selection (EVAL-SS): The EVAL-SS included all subjects who answered the self-selection question, probing question and follow-up questions (Part 1).
- Treated Set: Treated Set (TS): The TS included all subjects who self-selected to use the product, purchased the product, and then took at least one dose of drug (Part 2).
- FAS-AUS: Full Analysis Set for Actual Use Decision (FAS-AUS): The FAS-AUS included all subjects who self-selected to use the product, purchased the product, took at least one dose of drug and participated in at least 1 phone interview (Part 2).
Arm/Group | EVAL-SS | Treated Set | FAS-AUS
Serious Adverse Events (participants affected / at risk) | 10/679 | 10/351 | 9/321
Other Adverse Events (participants affected / at risk) | 26/679 | 26/351 | 22/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVAL-SS (N=679) | Treated Set (N=351) | FAS-AUS (N=321)
Abscess (Infections and infestations) | 1 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVAL-SS (N=679) | Treated Set (N=351) | FAS-AUS (N=321)
Nasopharyngitis (Infections and infestations) | 26 | 26 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.